CLINICAL TRIAL: NCT04672681
Title: Rehabilitation Including Structured Active Play for Preschoolers With Cancer.
Acronym: RePlay
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Danish Cancer Society (Other); Danish Child Cancer Foundation (Other); University of Copenhagen (Other)
Responsible Party: Principal Investigator, Hanne Baekgaard Larsen, Associate Professor, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RePlay-2020
Record Dates: First submitted 2020-12-03; First posted 2020-12-17 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Pediatric Cancer
Keywords: physical activity; preschool; cancer; play; social development; gross motor function
MeSH Terms: conditions — Neoplasms; Motor Activity

STUDY DESIGN:
Intervention Model Description: The intervention is a parallel model where the participants are randomized to either the intervention group or standard care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention group will receive a 6-month play-based physical activity intervention with daily play and movement activities starting from treatment initiation.
  Interventions: Behavioral: Play-based physical activity intervention
- Standard care (No Intervention): The control group will receive standard treatment and physiotherapy if needed.
  For ethical reasons, after the primary study end-point at six months, the participants and parents allocated to this group will be offered the same inspirational material and the possibility to participate in the group-based physical activity as the participants and parents allocated to the intervention group, but they will not receive education and supervision play-based physical activity with their child in the hospital room.

INTERVENTIONS:
Behavioral: Play-based physical activity intervention — The intervention group will participate in a six-month play-based physical activity intervention starting from their initiated treatment. The intervention combines hospital and home-based physical activity. Three days a week, there will be 45 minutes of group-based physical activity at the hospital during admissions or appointments at the outpatient clinic, supervised by an exercise professional or pediatric physiotherapist. Children who are isolated during treatment are offered supervised individual 45 min. training sessions 3 times a week as a substitute. During the other four days a week, or on days where the family is at home, the parents administer the play-based physical activity. At inclusion, the parents receive education and supervision on conducting play-based physical activity with their child in the hospital room or at home. They will receive inspiration material containing numerous different plays, games, and activities in different intensities.
  Arms: Intervention group

SUMMARY:
Treatment for childhood cancer causes treatment-related acute adverse events such as muscle weakness and physical incompetence. With long admissions, isolation, and long-term bed rest, this means reduced physical activity and, ultimately, gross motor functioning development is affected. Furthermore, the children participate less in sport and leisure activities, inhibiting social skills, and the children feel isolated from peers. The above makes it difficult for children to return to everyday activities. Physical activity in the form of play and movement activities is essential for preschool children's gross motor, social, and personal development- a development where parents play a crucial role.

Replay is a randomized controlled trial that will include 84 children with cancer aged 1-5 years at the University Hospital Copenhagen, Rigshospitalet. The children are included at the treatment initiation and are randomized to either the intervention group or the control group. The intervention consists of six months of daily structured play-based physical activity, including daily parent administered play and movement and three weekly group-based play and movement sessions at the hospital during admissions. Gross motor and physical function is measured with 1) Peabody Developmental Motor Scales, Second Edition (PDMS-2), Pediatric Evaluation of Disability Inventory (PEDI), Handgrip strength, and a six-minute walk test. The assessment time points are baseline (initiated timepoint), 3- and 6 months (endpoint) after initiated treatment. The intervention group will be observed and invited to participate in qualitative interviews. The control group will receive usual care and specific physiotherapy if needed.

DETAILED DESCRIPTION:
Aim

Project RePlay aims to investigate the effectiveness of a play-based physical activity intervention on gross motor functioning measured by Peabody Developmental Motor Scales, Second Edition (PDMS-2) with the primary end-point six months after diagnosis in children with newly diagnosed cancer aged 1-5 years old. The investigators hypothesize that the intervention will reduce short- and long-term physical and psychosocial consequences, including reduced gross motor function and lack of social interaction.

1. Background

   Physical play and movement activities are essential for preschool children's gross motor, social, and personal development. Through play and movement, children develop motor skills crucial for participation in physical and social activities throughout life. A study showed that an 18-week play intervention among healthy preschool children significantly improved (p<.0005) gross motor function in the intervention group compared with the control group. Play is also the children's first arena for socializing, and these interactions have an immense role in developing emotional, personal, and social skills. Physical play and movement activities are more than just physical exercise; it is social teamwork, emotions, and learning. Reduced physical activity or inactivity in children is highly dependent on three factors; 1) reduced dynapenia (muscle strength and power), 2) exercise deficit disorder (physical inactivity), and 3) physical illiteracy (reduced competence, confidence, and knowledge in movement). Due to more intensive treatment with chemotherapy, radiation, and surgery, children with cancer experience acute adverse events such as myopathy and neuropathy, resulting in muscle weakness, physical incompetence, and inactivity. Furthermore, treatment-related complications such as infections can cause extended periods of hospitalization, periods of isolation, and long-term bed rest. Thus, many children with cancer experience several physical side effects as impaired motor skills, physical capacity, and decreased motivation to engage in physical activity. The cancer treatment has a significant impact on the children's physical development and socialization as the lack of motor development leads to inactivity and less participation in sport and leisure activities. This leads to a reduced understanding of the social playing field in joint activities, and the children feel more isolated from peers. Children with cancer experiences challenges in all three factors leading to physical inactivity. Compared with siblings and the general population, these social and physical challenges persist for the rest of their lives. Hence, children diagnosed with cancer have lower school performance, lower education level, higher unemployment, and increased socioeconomic challenges. Thus, the investigators hypothesize that early initiated rehabilitation programs during initial treatment, focusing on maintaining a typical physical activity level, are crucial for continuing everyday activities during and after treatment.

   The rehabilitation, including social and physical activity and education in children and teenagers with cancer (RESPECT) study for children with cancer aged 6-18 years, showed that it is feasible to carry out physical tests and motivate them to participate in physical activities. Physical activity maintained the hospitalized children's physical fitness and gross motor function during treatment compared with hospitalized children who did not receive physical activity intervention. A systematic review covering international studies show similar findings; that physical activities positively affect mobility, physical fitness, muscle strength, and quality of life in children with cancer. Additionally, children with cancer who participate in structured physical activities during treatment have fewer admission days than children who received standard care, corresponding to a 17% reduction in hospitalization's total economic cost. Most studies focusing on physical activity as part of an early initiated rehabilitation program designed interventions for school children aged 6-18. Only a few of the studies include children under the age of 6 years. Each year 200 children and adolescents aged 0-18 years are diagnosed with cancer in Denmark. Of these, approximately one-third is diagnosed before the age of 5. None of the published studies on physical activity in pediatric oncology designed interventions for preschool children (1-5 years old). Thus, there is a lack of studies with an intervention designed for preschool children with cancer focusing on physical and social rehabilitation. Improvements in cure-rates of childhood cancer mean that today's 5-year survival is 85%. Thus, more research into the best strategies for physical activity and rehabilitation for all age groups of children with cancer is needed.

   A single study of parent-controlled physical activity at home included children with cancer from age 1-17. The intervention didn't improve the children's motor function compared with the control group, mainly due to poor adherence to the intervention. Project RESPECT shows that motivation and adherence to physical activity interventions are dependent on the support from "significant others" such as parents and exercise professionals. Parents are an essential resource for children with cancer. The parents follow the child's treatment closely, and the parents' support throughout the treatment is crucial for the child's need for presence and support so the child can feel safe and in control. Furthermore, the focus on home-based care is increasing to minimize hospital visits. Consequently, parents play an essential role in physical activity and rehabilitation for children with cancer. For preschool children, the parents' role is even more essential. When small children and parents play together, it creates a unique and safe environment where the children can be challenged physically and socially. Children's development is dependent on parents, and parents of a child with cancer must acquire the necessary skills concerning play and movement for the child.

   With project RePlay, the aim is to develop prophylactic strategies by investigating a play-based physical activity intervention for children with cancer aged 1-5 years to ensure the retention of natural motor and social development and participation in everyday activities. The hypothesis is that individual and social play and movement activities, with parents as resources, can reduce gross motor and social development impairments. Thus, the objectives of RePlay are:
   * To investigate the effects of a six-month play-based physical activity intervention in children with cancer, aged 1-5 years on gross motor function compared with a control group receiving usual care.
   * To investigate the children with cancer and the parents' experiences with a play-based physical activity intervention during treatment and the influence on the children's social and personal development.
2. Research plan

Design:

The randomized controlled trial study takes place at the Department of Pediatric Hematology/Oncology at Rigshospitalet. RePlay will include 84 children aged 1-5 years diagnosed with cancer. The children are randomized to either the intervention- or control group after the children have performed the baseline testing. The children will be stratified by age at inclusion (respectively, over and under three years old) and treatment group (hematologic malignancy, solid tumors, CNS-tumors). The intervention group will participate in a six-month play-based physical activity intervention starting from initiated treatment. The study will be an open-ended cohort where newly diagnosed patients are included on an ongoing basis.

The intervention will consist of 45 min daily play-based physical activities inspired by Mighty Moves from the study of Bellows et al. [5], where the activities are playful and focus on gross motor skills. The intervention combines hospital and home-based physical activity. Three days a week, there will be 45 minutes of group-based physical activity at the hospital for the children, siblings, and parents during admissions or appointments at the outpatient clinic. An exercise professional or pediatric physiotherapist administers the group-based sessions at the hospital. Children isolated in the hospital room are offered individual sessions as a substitute for the group-based sessions.

During the other four days a week or on days where the family is at home, the parents administer the play-based physical activity. The parents receive education and supervision on conducting play-based physical activity with their child in the hospital room or at home. The parents will receive inspiration material containing numerous different plays, games, and activities in different intensities, ensuring that their child is physically active every day with different intensity. The material is designed to engage the child in choosing what activities to do.

Due to age-specific development and movement, the children in the intervention group are split into two groups for the group-based sessions:

• Tumble: 1-2 years old • Tumble turbo: 3-5 years old

An example of a weekly schedule:

Monday: parent administered play

Tuesday: parents administered play OR group-based session at the hospital

Wednesday: parent administered play

Thursday: parents administered play OR group-based session at the hospital

Friday: parents administered play OR group-based session at the hospital

Saturday: parents administered play

Sunday: parents administered play

The control group will receive standard treatment and physiotherapy if needed. After six months of treatment, the child and parents will receive a status on the child's motor development and be invited to receive individual instructions and invited to participate in the social sessions.

Sample size:

Since there is no evidence on the potential effect of gross motor function in children with cancer, the sample size is estimated based on Bellows et al.'s (2013). The study objective was to research the potential of a play intervention on gross motor function in healthy preschool children measured by Peabody Developmental Motor Scales, Second Edition (PDMS-2). The sample size is estimated with an Alpha = 0,05 and Power = 80%. Based on a mean (SD) in the interventions group = 99,31 (9,07) and a mean (SD) in the control group = 93,24, n=70 (35 intervention group; 35 control group) are to be included. Assuming a 20% dropout rate, RePlay will include 84 children.

ELIGIBILITY:
Inclusion Criteria:

* Children diagnosed with cancer or benign disorders and are being treated with chemotherapy and/or radiation and are admitted to the Department of Pediatric Hematology/Oncology at University Hospital Copenhagen, Rigshospitalet.
* Children at the age of 1-5,9 years at diagnosis.
* Children whose parents can communicate in Danish.

Exclusion Criteria:

* Children with mental disabilities that complicates the ability to follow instructions.

Ages: 12 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 84 (Actual)
Dates: Start 2021-01-07 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Gross Motor Function | Baseline (treatment initiation)
  Gross Motor Function is measured with the gross motor function subscale of Peabody Developmental Motor Scales, Second Edition (PDMS-2). PDMS-2 gives a gross motor standard score summed by the standard score from the three gross motor domians; stationary, locomotion and object manipulation. The primary endpoint is after six months.
Gross Motor Function | 3 months after treatment initiation
  Gross Motor Function is measured with the gross motor function subscale of Peabody Developmental Motor Scales, Second Edition (PDMS-2). PDMS-2 gives a gross motor standard score summed by the standard score from the three gross motor domians; stationary, locomotion and object manipulation. The primary endpoint is after six months.
Gross Motor Function | 6 months after treatment initiation (primary endpoint)
  Gross Motor Function is measured with the gross motor function subscale of Peabody Developmental Motor Scales, Second Edition (PDMS-2). PDMS-2 gives a gross motor standard score summed by the standard score from the three gross motor domians; stationary, locomotion and object manipulation. The primary endpoint is after six months.
Gross Motor Function | 12 months after treatment initiation
  Gross Motor Function is measured with the gross motor function subscale of Peabody Developmental Motor Scales, Second Edition (PDMS-2). PDMS-2 gives a gross motor standard score summed by the standard score from the three gross motor domians; stationary, locomotion and object manipulation. The primary endpoint is after six months.
Gross Motor Function | 12 months after ended treatment
  Gross Motor Function is measured with the gross motor function subscale of Peabody Developmental Motor Scales, Second Edition (PDMS-2). PDMS-2 gives a gross motor standard score summed by the standard score from the three gross motor domians; stationary, locomotion and object manipulation. The primary endpoint is after six months.

SECONDARY OUTCOMES:
Level of child's function in everyday life | Baseline (treatment initiation)
  Level of function is measured through parent structured interviews with Pediatric Evaluation of Disability Inventory (PEDI) where parents answer wuestions about their child's function in three domains self-care, mobiliy and social functioning and the child's need for help in the same three domains. The primary endpoint is after six months.
Level of child's function in everyday life | 3 months after treatment initiation
  Level of function is measured through parent structured interviews with Pediatric Evaluation of Disability Inventory (PEDI) where parents answer wuestions about their child's function in three domains self-care, mobiliy and social functioning and the child's need for help in the same three domains. The primary endpoint is after six months.
Level of child's function in everyday life | 6 months after treatment initiation (primary endpoint)
  Level of function is measured through parent structured interviews with Pediatric Evaluation of Disability Inventory (PEDI) where parents answer wuestions about their child's function in three domains self-care, mobiliy and social functioning and the child's need for help in the same three domains. The primary endpoint is after six months.
Level of child's function in everyday life | 12 months after treatment initiation
  Level of function is measured through parent structured interviews with Pediatric Evaluation of Disability Inventory (PEDI) where parents answer wuestions about their child's function in three domains self-care, mobiliy and social functioning and the child's need for help in the same three domains. The primary endpoint is after six months.
Level of child's function in everyday life | 12 months after ended treatment
  Level of function is measured through parent structured interviews with Pediatric Evaluation of Disability Inventory (PEDI) where parents answer wuestions about their child's function in three domains self-care, mobiliy and social functioning and the child's need for help in the same three domains. The primary endpoint is after six months.
Handgrip strength | Baseline (treatment initiation)
  Handgrip strength measured with the KLS Martin Vigorimeter. Measures in bar. The primary endpoint is after six months.
Handgrip strength | 3 months after treatment initiation
  Handgrip strength measured with the KLS Martin Vigorimeter. Measures in bar. The primary endpoint is after six months.
Handgrip strength | 6 months after treatment initiation (primary endpoint)
  Handgrip strength measured with the KLS Martin Vigorimeter. Measures in bar. The primary endpoint is after six months.
Handgrip strength | 12 months after treatment initiation
  Handgrip strength measured with the KLS Martin Vigorimeter. Measures in bar. The primary endpoint is after six months.
Handgrip strength | 12 months after ended treatment
  Handgrip strength measured with the KLS Martin Vigorimeter. Measures in bar. The primary endpoint is after six months.
Six-minute walk | Baseline (treatment initiation)
  Six-minute walk test is done with the measurement of total meters walk after 6 minutes. The primary endpoint is after six months.
Six-minute walk | 3 months after treatment initiation
  Six-minute walk test is done with the measurement of total meters walk after 6 minutes. The primary endpoint is after six months.
Six-minute walk | 6 months after treatment initiation (primary endpoint)
  Six-minute walk test is done with the measurement of total meters walk after 6 minutes. The primary endpoint is after six months.
Six-minute walk | 12 months after treatment initiation
  Six-minute walk test is done with the measurement of total meters walk after 6 minutes. The primary endpoint is after six months.
Six-minute walk | 12 months after ended treatment
  Six-minute walk test is done with the measurement of total meters walk after 6 minutes. The primary endpoint is after six months.
Two-minute walk | Baseline (treatment initiation)
  Two-minute walk test is done with the measurement of total meters walk after 2 minutes during the six-minute walk. The primary endpoint is after six months.
Two-minute walk | 3 months after treatment initiation
  Two-minute walk test is done with the measurement of total meters walk after 2 minutes during the six-minute walk. The primary endpoint is after six months.
Two-minute walk | 6 months after treatment initiation (primary endpoint)
  Two-minute walk test is done with the measurement of total meters walk after 2 minutes during the six-minute walk. The primary endpoint is after six months.
Two-minute walk | 12 months after treatment initiation
  Two-minute walk test is done with the measurement of total meters walk after 2 minutes during the six-minute walk. The primary endpoint is after six months.
Two-minute walk | 12 months after ended treatment
  Two-minute walk test is done with the measurement of total meters walk after 2 minutes during the six-minute walk. The primary endpoint is after six months.

OTHER OUTCOMES:
Child's health-related quality of life - Generic Core Scale | Baseline (treatment initiation)
  PedsQl Generic Core Scale - Proxy. Parents answer the questions about their child's helths-related quality of life. The primary endpoint is after six months.
Child's health-related quality of life - Generic Core Scale | 6 months after treatment initiation (primary endpoint)
  PedsQl Generic Core Scale - Proxy. Parents answer the questions about their child's helths-related quality of life. The primary endpoint is after six months.
Child's health-related quality of life - Generic Core Scale | 12 months after treatment initiation
  PedsQl Generic Core Scale - Proxy. Parents answer the questions about their child's helths-related quality of life. The primary endpoint is after six months.
Child's health-related quality of life - Generic Core Scale | 12 months after ended treatment
  PedsQl Generic Core Scale - Proxy. Parents answer the questions about their child's helths-related quality of life. The primary endpoint is after six months.
Child's health-related quality of life - Cancer | Baseline (treatment initiation)
  PedsQl Cancer - Proxy. Parents answer the questions about their child's helths-related quality of life. The primary endpoint is after six months.
Child's health-related quality of life - Cancer | 6 months after treatment initiation (primary endpoint)
  PedsQl Cancer - Proxy. Parents answer the questions about their child's helths-related quality of life. The primary endpoint is after six months.
Child's health-related quality of life - Fatigue Scale | Baseline (treatment initiation)
  PedsQl Fatigue Scale - Proxy. Parents answer the questions about their child's helths-related quality of life. The primary endpoint is after six months.
Child's health-related quality of life - Fatigue Scale | 6 months after treatment initiation (primary endpoint)
  PedsQl Fatigue Scale - Proxy. Parents answer the questions about their child's helths-related quality of life. The primary endpoint is after six months.
Child's health-related quality of life - Fatigue Scale | 12 months after treatment initiation
  PedsQl Fatigue Scale - Proxy. Parents answer the questions about their child's helths-related quality of life. The primary endpoint is after six months.
Child's health-related quality of life - Fatigue Scale | 12 months after ended treatment
  PedsQl Fatigue Scale - Proxy. Parents answer the questions about their child's helths-related quality of life. The primary endpoint is after six months.
Parents health-related quality of life | Baseline (treatment initiation)
  36-Item Short Form Survey Instrument (SF 36). Parents answer questions about their own health-related quality of life. The primary endpoint is after six months.
Parents health-related quality of life | 6 months after treatment initiation (primary endpoint)
  36-Item Short Form Survey Instrument (SF 36). Parents answer questions about their own health-related quality of life. The primary endpoint is after six months.
Parents health-related quality of life | 12 months after treatment initiation
  36-Item Short Form Survey Instrument (SF 36). Parents answer questions about their own health-related quality of life. The primary endpoint is after six months.
Parents health-related quality of life | 12 months after ended treatment
  36-Item Short Form Survey Instrument (SF 36). Parents answer questions about their own health-related quality of life. The primary endpoint is after six months.
Semi-structured interviews and observations | Baseline (treatment initiation) and 6 months.
  We expect to conduct additional studies that will include empirical data collected through semi-structured interviews and observations. The empirical data collected will be analyzed and reported in separate articles.
  The children and the parents in the intervention group will be interviewed (children with no language; only the parents are interviewed). The interview is done pre-and post-intervention. Observational fieldwork will be carried out during the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Hanne B Larsen, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bjorklund DF, Brown RD. Physical play and cognitive development: integrating activity, cognition, and education. Child Dev. 1998 Jun;69(3):604-6. PMID 9680673
- [Background] Bellows LL, Davies PL, Anderson J, Kennedy C. Effectiveness of a physical activity intervention for Head Start preschoolers: a randomized intervention study. Am J Occup Ther. 2013 Jan-Feb;67(1):28-36. doi: 10.5014/ajot.2013.005777. PMID 23245780
- [Background] Faigenbaum AD, Rebullido TR, MacDonald JP. Pediatric Inactivity Triad: A Risky PIT. Curr Sports Med Rep. 2018 Feb;17(2):45-47. doi: 10.1249/JSR.0000000000000450. No abstract available. PMID 29420346
- [Background] Gatta G, Zigon G, Capocaccia R, Coebergh JW, Desandes E, Kaatsch P, Pastore G, Peris-Bonet R, Stiller CA; EUROCARE Working Group. Survival of European children and young adults with cancer diagnosed 1995-2002. Eur J Cancer. 2009 Apr;45(6):992-1005. doi: 10.1016/j.ejca.2008.11.042. Epub 2009 Feb 21. PMID 19231160
- [Background] Smith MA, Seibel NL, Altekruse SF, Ries LA, Melbert DL, O'Leary M, Smith FO, Reaman GH. Outcomes for children and adolescents with cancer: challenges for the twenty-first century. J Clin Oncol. 2010 May 20;28(15):2625-34. doi: 10.1200/JCO.2009.27.0421. Epub 2010 Apr 19. PMID 20404250
- [Background] Gibson TM, Mostoufi-Moab S, Stratton KL, Leisenring WM, Barnea D, Chow EJ, Donaldson SS, Howell RM, Hudson MM, Mahajan A, Nathan PC, Ness KK, Sklar CA, Tonorezos ES, Weldon CB, Wells EM, Yasui Y, Armstrong GT, Robison LL, Oeffinger KC. Temporal patterns in the risk of chronic health conditions in survivors of childhood cancer diagnosed 1970-99: a report from the Childhood Cancer Survivor Study cohort. Lancet Oncol. 2018 Dec;19(12):1590-1601. doi: 10.1016/S1470-2045(18)30537-0. Epub 2018 Nov 8. PMID 30416076
- [Background] Ness KK, Kaste SC, Zhu L, Pui CH, Jeha S, Nathan PC, Inaba H, Wasilewski-Masker K, Shah D, Wells RJ, Karlage RE, Robison LL, Cox CL. Skeletal, neuromuscular and fitness impairments among children with newly diagnosed acute lymphoblastic leukemia. Leuk Lymphoma. 2015 Apr;56(4):1004-11. doi: 10.3109/10428194.2014.944519. Epub 2014 Aug 20. PMID 25030039
- [Background] Thorsteinsson T, Larsen HB, Schmiegelow K, Thing LF, Krustrup P, Pedersen MT, Christensen KB, Mogensen PR, Helms AS, Andersen LB. Cardiorespiratory fitness and physical function in children with cancer from diagnosis throughout treatment. BMJ Open Sport Exerc Med. 2017 May 12;3(1):e000179. doi: 10.1136/bmjsem-2016-000179. eCollection 2017. PMID 28761697
- [Background] Darcy L, Enskar K, Bjork M. Young children's experiences of living an everyday life with cancer - A three year interview study. Eur J Oncol Nurs. 2019 Apr;39:1-9. doi: 10.1016/j.ejon.2018.12.007. Epub 2018 Dec 23. PMID 30850132
- [Background] Hildenbrand AK, Clawson KJ, Alderfer MA, Marsac ML. Coping with pediatric cancer: strategies employed by children and their parents to manage cancer-related stressors during treatment. J Pediatr Oncol Nurs. 2011 Nov-Dec;28(6):344-54. doi: 10.1177/1043454211430823. PMID 22194147
- [Background] Bjork M, Nordstrom B, Hallstrom I. Needs of young children with cancer during their initial hospitalization: an observational study. J Pediatr Oncol Nurs. 2006 Jul-Aug;23(4):210-9. doi: 10.1177/1043454206289737. PMID 16766686
- [Background] Gibson F, Aldiss S, Horstman M, Kumpunen S, Richardson A. Children and young people's experiences of cancer care: a qualitative research study using participatory methods. Int J Nurs Stud. 2010 Nov;47(11):1397-407. doi: 10.1016/j.ijnurstu.2010.03.019. Epub 2010 Apr 28. PMID 20430388
- [Background] Vannatta K, Gerhardt CA, Wells RJ, Noll RB. Intensity of CNS treatment for pediatric cancer: prediction of social outcomes in survivors. Pediatr Blood Cancer. 2007 Oct 15;49(5):716-22. doi: 10.1002/pbc.21062. PMID 17096410
- [Background] Almqvist L, Hellnas P, Stefansson M, Granlund M. 'I can play!' young children's perceptions of health. Pediatr Rehabil. 2006 Jul-Sep;9(3):275-84. doi: 10.1080/13638490500521303. PMID 17050405
- [Background] van Brussel M, Takken T, van der Net J, Engelbert RH, Bierings M, Schoenmakers MA, Helders PJ. Physical function and fitness in long-term survivors of childhood leukaemia. Pediatr Rehabil. 2006 Jul-Sep;9(3):267-74. doi: 10.1080/13638490500523150. PMID 17050404
- [Background] Ness KK, Baker KS, Dengel DR, Youngren N, Sibley S, Mertens AC, Gurney JG. Body composition, muscle strength deficits and mobility limitations in adult survivors of childhood acute lymphoblastic leukemia. Pediatr Blood Cancer. 2007 Dec;49(7):975-81. doi: 10.1002/pbc.21091. PMID 17091482
- [Background] Ness KK, Hudson MM, Pui CH, Green DM, Krull KR, Huang TT, Robison LL, Morris EB. Neuromuscular impairments in adult survivors of childhood acute lymphoblastic leukemia: associations with physical performance and chemotherapy doses. Cancer. 2012 Feb 1;118(3):828-38. doi: 10.1002/cncr.26337. Epub 2011 Jul 15. PMID 21766297
- [Background] Frederiksen LE, Mader L, Feychting M, Mogensen H, Madanat-Harjuoja L, Malila N, Tolkkinen A, Hasle H, Winther JF, Erdmann F. Surviving childhood cancer: a systematic review of studies on risk and determinants of adverse socioeconomic outcomes. Int J Cancer. 2019 Apr 15;144(8):1796-1823. doi: 10.1002/ijc.31789. Epub 2018 Oct 30. PMID 30098012
- [Background] Nielsen MKF, Christensen JF, Frandsen TL, Thorsteinsson T, Andersen LB, Christensen KB, Nersting J, Faber M, Schmiegelow K, Larsen HB. Testing physical function in children undergoing intense cancer treatment-a RESPECT feasibility study. Pediatr Blood Cancer. 2018 Aug;65(8):e27100. doi: 10.1002/pbc.27100. Epub 2018 May 9. PMID 29741279
- [Background] Braam KI, van der Torre P, Takken T, Veening MA, van Dulmen-den Broeder E, Kaspers GJ. Physical exercise training interventions for children and young adults during and after treatment for childhood cancer. Cochrane Database Syst Rev. 2016 Mar 31;3(3):CD008796. doi: 10.1002/14651858.CD008796.pub3. PMID 27030386
- [Background] Morales JS, Santana-Sosa E, Santos-Lozano A, Bano-Rodrigo A, Valenzuela PL, Rincon-Castanedo C, Fernandez-Moreno D, Gonzalez Vicent M, Perez-Somarriba M, Madero L, Lassaletta A, Fiuza-Luces C, Lucia A. Inhospital exercise benefits in childhood cancer: A prospective cohort study. Scand J Med Sci Sports. 2020 Jan;30(1):126-134. doi: 10.1111/sms.13545. Epub 2019 Oct 6. PMID 31482597
- [Background] Hartman A, te Winkel ML, van Beek RD, de Muinck Keizer-Schrama SM, Kemper HC, Hop WC, van den Heuvel-Eibrink MM, Pieters R. A randomized trial investigating an exercise program to prevent reduction of bone mineral density and impairment of motor performance during treatment for childhood acute lymphoblastic leukemia. Pediatr Blood Cancer. 2009 Jul;53(1):64-71. doi: 10.1002/pbc.21942. PMID 19283791
- [Background] Thorsteinsson T, Schmiegelow K, Thing LF, Andersen LB, Helms AS, Ingersgaard MV, Lindgren LH, Larsen HB. Classmates motivate childhood cancer patients to participate in physical activity during treatment: A qualitative study. Eur J Cancer Care (Engl). 2019 Sep;28(5):e13121. doi: 10.1111/ecc.13121. Epub 2019 Jun 18. PMID 31215079
- [Background] Hansson H, Kjaergaard H, Schmiegelow K, Hallstrom I. Hospital-based home care for children with cancer: a qualitative exploration of family members' experiences in Denmark. Eur J Cancer Care (Engl). 2012 Jan;21(1):59-66. doi: 10.1111/j.1365-2354.2011.01280.x. Epub 2011 Aug 18. PMID 21848580
- [Background] Hansson H, Hallstrom I, Kjaergaard H, Johansen C, Schmiegelow K. Hospital-based home care for children with cancer. Pediatr Blood Cancer. 2011 Sep;57(3):369-77. doi: 10.1002/pbc.23047. Epub 2011 May 18. PMID 21594980
- [Background] Schroder H, Rechnitzer C, Wehner PS, Rosthoj S, Moller JK, Lausen B, Petersen G, Norgaard M. Danish Childhood Cancer Registry. Clin Epidemiol. 2016 Oct 25;8:461-464. doi: 10.2147/CLEP.S99508. eCollection 2016. PMID 27822085
- [Background] Stahlhut M, Christensen J, Aadahl M. Applicability and intrarespondent reliability of the pediatric evaluation of disability inventory in a random Danish sample. Pediatr Phys Ther. 2010 Summer;22(2):161-9. doi: 10.1097/PEP.0b013e3181dbf965. PMID 20473099
- [Background] Hager-Ross C, Rosblad B. Norms for grip strength in children aged 4-16 years. Acta Paediatr. 2002;91(6):617-25. doi: 10.1080/080352502760068990. PMID 12162590
- [Background] Enright PL. The six-minute walk test. Respir Care. 2003 Aug;48(8):783-5. PMID 12890299
- [Background] Robertson A, Deitz J. A description of grip strength in preschool children. Am J Occup Ther. 1988 Oct;42(10):647-52. doi: 10.5014/ajot.42.10.647. PMID 3202109
- [Background] Neumann S, Kwisda S, Krettek C, Gaulke R. Comparison of the Grip Strength Using the Martin-Vigorimeter and the JAMAR-Dynamometer: Establishment of Normal Values. In Vivo. 2017 Sep-Oct;31(5):917-924. doi: 10.21873/invivo.11147. PMID 28882959
- [Derived] Pouplier A, Fridh MK, Christensen J, Hoyer A, Schmidt-Andersen P, Winther H, Larsen HB. Rehabilitation including structured active play intervention for preschoolers with cancer during treatment: A RePlay qualitative study of parents' experiences. Eur J Oncol Nurs. 2024 Aug;71:102639. doi: 10.1016/j.ejon.2024.102639. Epub 2024 Jun 7. PMID 38878692
- [Derived] Pouplier A, Fridh MK, Christensen J, Ruiz-Molsgaard H, Hoyer A, Schmidt-Andersen P, Winther H, Larsen HB. The potential of structured active play for social and personal development in preschoolers during cancer treatment: A qualitative RePlay study. J Adv Nurs. 2024 Apr;80(4):1607-1618. doi: 10.1111/jan.15923. Epub 2023 Nov 10. PMID 37950393
- [Derived] Pouplier A, Winther H, Christensen J, Schmidt-Andersen P, Zhang H, Frandsen TL, Schmiegelow K, Fridh MK, Larsen HB. Rehabilitation Including Structured Active Play for Preschoolers With Cancer (RePlay)-Study Protocol for a Randomized Controlled Trial. Front Pediatr. 2022 May 9;10:834512. doi: 10.3389/fped.2022.834512. eCollection 2022. PMID 35615627

DOCUMENTS (1):
  • Statistical Analysis Plan (2021-10-08): https://cdn.clinicaltrials.gov/large-docs/81/NCT04672681/SAP_000.pdf